CLINICAL TRIAL: NCT00957684
Title: Efficacy and Safety of Eslicarbazepine Acetate (BIA 2-093) as Adjunctive Therapy for Refractory Partial Seizures in a Double-blind, Randomised, Placebo-controlled, Parallel-group, Multicentre Clinical Trial.
Brief Title: Efficacy and Safety of Eslicarbazepine Acetate as Adjunctive Therapy for Refractory Partial Seizures
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bial - Portela C S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BIA-2093-301
Record Dates: First submitted 2009-08-10; First posted 2009-08-12 (Estimated); Results first posted 2013-10-10 (Estimated); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Refractory Partial Epilepsy
Keywords: refractory; partial; epilepsy
MeSH Terms: conditions — Epilepsies, Partial; Epilepsy | interventions — eslicarbazepine acetate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- ESL 400 mg once daily (Experimental): ESL was supplied in 400-mg and 800-mg tablets
  Interventions: Drug: eslicarbazepine acetate
- ESL 800 mg once daily (Experimental): ESL was supplied in 400-mg and 800-mg tablets
  Interventions: Drug: eslicarbazepine acetate
- ESL 1200 mg once daily (Experimental): ESL was supplied in 400-mg and 800-mg tablets
  Interventions: Drug: eslicarbazepine acetate
- placebo (Placebo Comparator): Placebo matching tablets
  Interventions: Drug: placebo
- ESL - PART II (Experimental): During Part II of the study all patients received Eslicarbazepine Acetate (ESL), including those who had been treated with placebo during Part I. ESL was supplied as scored 800 mg tablets; once daily administration by oral route.
  Interventions: Drug: eslicarbazepine acetate

INTERVENTIONS:
Drug: eslicarbazepine acetate — once-daily oral tablet
  Other Names: Zebinix
  Arms: ESL - PART II; ESL 1200 mg once daily; ESL 400 mg once daily; ESL 800 mg once daily
Drug: placebo — once daily placebo comparator
  Arms: placebo

SUMMARY:
This was a phase III 4-part study in multiple centres. Part I was a 26-week parallel-group, randomised, placebo-controlled period (8 weeks single-blind placebo baseline, 2 weeks double-blind titration, 12 weeks maintenance, and 4 weeks tapering off). After completing the baseline period, patients were randomised in a 1:1:1:1 ratio to 1 of 3 ESL dose levels or to placebo. Part II was a 1-year open-label extension for patients who had completed Part I. The starting dose was 800 mg once daily and could be titrated up or down at 400-mg intervals between 400 and 1200 mg. Part III was an additional 1-year open-label extension for patients who had completed Part II, had participated in the post-Part II study extension, which allowed patients to continue treatment with ESL, or had continued to take ESL in a compassionate use program. ESL starting doses were the same as received at the end of Part II, during post-Part II study extension, or under compassionate use, and could be titrated up or down at 400-mg intervals between 400 and 1200 mg once daily. Part IV was a study extension to allow patients to continue ESL treatment after the end of Part III until marketing authorisation or discontinuation of clinical development.

DETAILED DESCRIPTION:
Duration of Treatment: The duration of Part I was 26 weeks: 8 weeks of placebo run-in, 2 weeks of dose titration, 12 weeks of maintenance, and 4 weeks of tapering-off period. The duration of Part II was 1 year. The duration of Part III was planned to be 1 year (some patients were treated for >1 year). The duration of Part IV was >3 years (patients could continue treatment with ESL until market availability).

ELIGIBILITY:
Inclusion Criteria:

* written informed consent signed by patient
* aged 18 years or more
* documented diagnosis of simple or complex partial seizures with or without secondary generalisation since at least 12 months prior to screening
* at least 4 partial seizures in each 4 week period during the last 8 weeks prior to screening, currently treated with 1 or 2 AEDs (any except oxcarbazepine and felbamate), in a stable dose regimen during at least 2 months prior to screening (patients using vigabatrin should have been on this medication for at least 1 year with no deficit in visual field identified)
* excepting epilepsy, patient is judged to be in general good health based on medical history, physical examination and laboratory tests
* post-menopausal or otherwise incapable of becoming pregnant by reason of surgery or tubal ligation; in case of woman of childbearing potential, patient must present a serum beta-hCG test consistent with a non-gravid state and agree to remain abstinent or use reliable contraception (oral contraception should be combined with a barrier method)

Exclusion Criteria:

* only simple partial seizures with no motor symptomatology (classified as A2-4 according to the International Classification of Epileptic Seizures) that are not video-EEG documented
* primarily generalised epilepsy
* known rapid progressive neurological disorder; history of status epilepticus or cluster seizures (i.e., 3 or more seizures within 30 minutes) within the 3 months prior to screening
* seizures of psychogenic origin within the last 2 years
* history of schizophrenia or suicide attempt
* currently on or with exposure to felbamate or oxcarbazepine more within one month of screening
* using benzodiazepines on more than on an occasional basis (except when used chronically as AED)
* previous use of ESL or participation in a clinical study with ESL
* known hypersensitivity to carbamazepine, oxcarbazepine or chemically related substances
* history of abuse of alcohol, drugs or medications within the last 2 years
* uncontrolled cardiac, renal, hepatic, endocrine, gastrointestinal, metabolic, haematological or oncology disorder
* second or third-degree atrioventricular blockade not corrected with a pacemaker
* relevant clinical laboratory abnormalities

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 402 (Actual)
Dates: Start 2004-07; Primary Completion 2005-11 (Actual); Study Completion 2007-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Christian Elger, Principal Investigator — Department of Epileptology, Friedrich Wilhelms University Bonn; Prof. Peter Halasz, Principal Investigator — National Institute of Psychiatry and Neurology, Budapest, Hungary
Locations (1):
- Bial - Portela & Cª, S.A., São Mamede do Coronado, Portugal

REFERENCES:
- [Derived] Andermann E, Rosenfeld W, Penovich P, Rogin J, Cendes F, Carreno M, Ramsay RE, Ben-Menachem E, Gama H, Rocha F, Soares-da-Silva P, Tosiello R, Blum D, Grinnell T. Comparative analysis of the safety and tolerability of eslicarbazepine acetate in older (>/=60 years) and younger (18-59 years) adults. Epilepsy Res. 2021 Jan;169:106478. doi: 10.1016/j.eplepsyres.2020.106478. Epub 2020 Oct 10. PMID 33338829

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study initiation date: 15/July/2004(first visit of the first patient) Study Part I completion date: 09/November/2005(last Part I visit of the last patient) Study Part II initiation date: 11 JAN 2005 (first Part II visit of the first patient) Study Part II completion date: 04 JAN 2007 (last Part II visit of the last patient)
Pre-assignment Details: After completing the baseline period, patients were randomised in a 1:1:1:1 ratio to 1 of the 3 Eslicarbazepine acetate (ESL) dose levels or to placebo.
  Part II was a 1-year open-label extension for patients who had completed Part I
Groups:
- ESL 1200 mg Once Daily; ESL 800 mg Once Daily; ESL 400 mg Once Daily: eslicarbazepine acetate : once-daily oral tablet
- Placebo: placebo : once daily placebo comparator
- ESL - Part II: During Part II of the study all patients received ESL, including those who had been treated with placebo during Part I. The duration of treatment during Part II was one year for all patients completing the study.
Period: PART I
Arm/Group | ESL 1200 mg Once Daily | ESL 800 mg Once Daily | ESL 400 mg Once Daily | Placebo | ESL - Part II
Started | 102 | 98 | 100 | 102 | 0
Randomised (Safety Population) | 102 | 98 | 100 | 102 | 0
Intention-to-treat (ITT) Population | 98 | 98 | 99 | 102 | 0
Per-protocol (PP)Population | 72 | 86 | 94 | 91 | 0
Completed | 71 | 85 | 90 | 84 | 0
Not Completed | 31 | 13 | 10 | 18 | 0
Period: PART II
Arm/Group | ESL 1200 mg Once Daily | ESL 800 mg Once Daily | ESL 400 mg Once Daily | Placebo | ESL - Part II
Started | 0 | 0 | 0 | 0 | 314
Patients Entered Part II | 0 | 0 | 0 | 0 | 314
Completed | 0 | 0 | 0 | 0 | 239
Not Completed | 0 | 0 | 0 | 0 | 75

BASELINE CHARACTERISTICS:
Groups:
- ESL 1200 mg: 400-mg + 800-mg; once daily administration by oral route
- ESL 800 mg: 800-mg; once daily administration by oral route
- ESL 400 mg: 400-mg; once daily administration by oral route
- Placebo: Placebo tablets; once daily administration by oral route
- Total: Total of all reporting groups
Arm/Group | ESL 1200 mg | ESL 800 mg | ESL 400 mg | Placebo | Total
Number analyzed (Participants) | 102 | 98 | 100 | 102 | 402
Age, Customized [Number; unit: participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 70 years | 102 | 96 | 99 | 102 | 399
  >70 years | 0 | 2 | 1 | 0 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 57 | 44 | 49 | 54 | 204
  Male | 45 | 54 | 51 | 48 | 198

OUTCOME MEASURES:

1. Primary Outcome: Part I: Seizure Frequency
Description: The primary efficacy endpoint is the natural log transformation of the seizure frequency per 4 weeks. The primary efficacy analysis was based on the intention-to-treat (ITT) population. Efficacy analyses were performed chiefly using data from the 12-week maintenance period in Part I of the study. The primary efficacy variable is the ln transformation of the seizure frequency per 4 weeks. Seizure frequency was compared between each active treatment group and the placebo group using an ANCOVA that models seizure frequency as a function of baseline seizure frequency and treatment.to a "frequency per 4 weeks" basis
Time Frame: 12-week maintenance period
Population: The primary efficacy analysis was based on the ITT population.
Measure: Least Squares Mean (95% Confidence Interval); unit: ln (Seizures) per 4 weeks
Groups:
- Placebo: Placebo tablets matching the 400-mg and 800-mg active substance tablets were supplied; once daily administration by oral route.
- ESL 400 mg: ESL was supplied in 400-mg tablets; once daily administration by oral route.
- ESL 800 mg: ESL was supplied in 800-mg tablets; once daily administration by oral route.
- ESL 1200 mg: ESL was supplied in 400-mg and 800-mg tablets; once daily administration by oral route.
Arm/Group | Placebo | ESL 400 mg | ESL 800 mg | ESL 1200 mg
Number analyzed (Participants) | 102 | 99 | 98 | 98
ln (Seizures) per 4 weeks | 7.64 (0.0563) [6.78 to 8.58] | 6.73 (0.0563) [5.93 to 7.60] | 5.66 (0.0558) [4.92 to 6.45] | 5.35 [4.63 to 6.12]

ADVERSE EVENTS:
Time Frame: 26-week
Description: Safety endpoints included Adverse events (AEs), clinical laboratory tests (haematology, coagulation, biochemistry, thyroid function, and urinalysis), vital signs and weight, electrocardiogram, and blood trough levels of concomitant Anti-epileptic drug (AEDs).
Arm/Group | ESL 1200 mg Once Daily | ESL 400 mg Once Daily | ESL 800 mg Once Daily | Placebo
Serious Adverse Events (participants affected / at risk) | 3/102 | 9/100 | 4/98 | 3/102
Other Adverse Events (participants affected / at risk) | 62/102 | 27/100 | 49/98 | 14/102
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | ESL 1200 mg Once Daily (N=102) | ESL 400 mg Once Daily (N=100) | ESL 800 mg Once Daily (N=98) | Placebo (N=102)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Angina pectoris (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Asthenia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Death (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dental caries (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Drug toxicity (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lower limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Traumatic brain injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pseudarthrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ataxia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Convulsion (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0/0 (0) | 1 (1) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Exanthem (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ESL 1200 mg Once Daily (N=102) | ESL 400 mg Once Daily (N=100) | ESL 800 mg Once Daily (N=98) | Placebo (N=102)
Dizziness (Nervous system disorders) | 14 (14) | 4 (4) | 14 (14) | 2 (2)
Headache (Nervous system disorders) | 11 (11) | 5 (5) | 9 (9) | 6 (6)
Somnolence (Nervous system disorders) | 10 (10) | 6 (6) | 9 (9) | 2 (2)
Diplopia (Eye disorders) | 11 (11) | 2 (2) | 7 (7) | 0 (0)
Nausea (Gastrointestinal disorders) | 5 (5) | 2 (2) | 4 (4) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 6 (6) | 2 (2) | 2 (2) | 1 (1)
Influenza (Infections and infestations) | 4 (4) | 3 (3) | 4 (4) | 0 (0)
Complex partial seizures (Nervous system disorders) | 3 (3) | 3 (3) | 1 (1) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other